CLINICAL TRIAL: NCT02487277
Title: Perioperative Stromal Depletion Strategies in Pancreatic Ductal Adenocarcinoma
Brief Title: PEGPH20, Gemicitabine and Nab-Paclitaxel for Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Andrew Ko (Other)
Responsible Party: Sponsor-Investigator, Andrew Ko, Professor of Clinical Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144515; NCI-2015-01213 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Adenocarcinoma
Keywords: Pancreatic
MeSH Terms: conditions — Adenocarcinoma | interventions — PEGPH20; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination therapy with 1 week Run-In (Experimental): PEGPH20: 3ug/kg on Days 1 and 4
  1 cycle = 28 days
  PEGPH20: 3ug/kg on Days 1, 8, 15
  Gemcitabine: 1000mg/m^2 on Days 1, 8, 15
  Nab-paclitaxel: 125mg/m^2 on Days 1, 8, 15
  Interventions: Drug: PEGPH20; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Combination therapy alone (Experimental): 1 cycle = 28 days
  PEGPH20: 3ug/kg on Days 1, 8, 15
  Gemcitabine: 1000mg/m^2 on Days 1, 8, 15
  Nab-paclitaxel: 125mg/m^2 on Days 1, 8, 15
  Interventions: Drug: PEGPH20; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: PEGPH20
Drug: Gemcitabine
Drug: Nab-paclitaxel

SUMMARY:
We will be conducting a Phase II study investigating PEGPH20 in combination with gemcitabine and nab-paclitaxel in patients with borderline resectable pancreatic ductal adenocarcinoma (PDAC) at the Helen Diller Family Comprehensive Cancer Center at University of California, San Francisco (UCSF). There are multiple definitions of borderline resectable PDAC including the MD Anderson definition and the criteria developed during the Consensus Conference sponsored by the American Hepato-Pancreato-Biliary Association, Society of Surgical Oncology, and Society for Surgery of the Alimentary Tract. Borderline resectable PDAC cases will be identified per the definition developed in the currently running inter-group pilot trial for borderline resectable pancreatic cancer (NCT01821612). Per this trial, borderline resectable PDAC is defined as "presence of any one or more of the following on CT:

* An interface between the primary tumor and the superior mesenteric vein or portal vein (SMV-PV) measuring ≥ 180° of the circumference of the vessel wall
* Short-segment occlusion of the SMV-PV with normal vein above and below the level of obstruction that is amenable to resection and venous reconstruction
* Short segment interface (of any degree) between tumor and hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and reconstruction.
* An interface between the tumor, and Superior mesenteric artery (SMA) measuring < 180º of the circumference of the vessel wall.

This trial will be conducted in two parts. In Part I, pre-treatment endoscopic ultrasound (EUS)-guided core biopsies of the pancreatic tumor, CA 19-9 levels and functional MRIs including Dynamic contrast-enhanced (DCE)-MRI and Diffusion-weighted magnetic resonance imaging (DWI-MRI) will be obtained for the first fifteen patients enrolled. After a 1-week run-in period with PEGPH20 on days 1 and 4, patients will have repeat EUS-guided core biopsies, functional MRI, CA 19-9 level and baseline CT chest, abdomen and pelvis. Subsequently, patients will be started on treatment with PEGPH20, gemcitabine and nab-paclitaxel given weekly for 3 weeks, every 28 days. To evaluate the disease response to treatment, CA 19-9 levels will be checked monthly and restaging CT chest, abdomen and pelvis will be obtained every 8 weeks. If there is disease progression at any point in the study, patients will be taken off of study and alternative treatments will be offered. At the completion of 4 cycles of therapy, restaging CT scans will be obtained to determine resectability. If the patients are found to have resectable disease, an additional functional MRI will be obtained to evaluate the PDAC stroma. If the patients are able to have successful surgeries, tissue analyses will be performed on the resected pancreatic tumor. These patients will then proceed to get 2 cycles of adjuvant chemotherapy with gemcitabine and nab-paclitaxel. If the patients are deemed to be surgical candidates but are found to have unresectable disease in the operating room, an intraoperative core biopsy of the pancreatic tumor will be obtained for tissue analyses. At the time of initiation of therapy with PEGPH20, patients will be started on prophylactic dose of enoxaparin 1 mg/kg subcutaneous daily. This will be continued throughout the study participation.

In Part II, an additional 21 patients will be enrolled, and will begin neoadjuvant therapy with PEGPH20, gemcitabine and nab-paclitaxel without the 1 week run-in of PEGPH20-only or the pre- and post-run-in EUS-guided biopsies.

DETAILED DESCRIPTION:
For Specific Aim 1, we will be monitoring the post-operative complication of clinically relevant pancreatic fistula within one week of surgery per the standard clinical guidelines as noted above. Common clinical presentations of pancreatic fistula include abdominal pain, leukocytosis and fever (temperature >100.4 degrees). Diagnostic work-up of pancreatic fistula will be with CT abdomen with contrast, which has a sensitivity of 63% and specificity of 83% for detecting pancreatic fistula. The pancreatic fistulas will be categorized into grades A, B or C as previously reported. Our study will be investigating only clinically relevant pancreatic fistulas, i.e. grades B or C. Depending on the grade of pancreatic fistula, patients will be treated as indicated with conservative treatment options including bowel rest, antibiotics, somatostatin analogues and percutaneous drainage or surgical re-exploration. We will also track other relevant post-operative complications such as delayed wound healing, development of wound dehiscence or wound infection.

The tissue analyses will include review of the immunohistochemical (IHC) stains for actin, hyaluronic acid staining with binding protein probe, proliferation as measured by ki-67% and Phospho-histone H3 (Ph-H3); cell apoptosis as evaluated by IHC stain for cleaved caspase 3 (CC3) and Tunel. If limited tissue sample is obtained via the core biopsies, the priority of tissue analysis will be as follows: (1) fixed in formalin for H&E and IHC (Ph-H3; CC3/Tunel; Hyaluronic Acid (HA) binding); (2) fixed in Optimal Cutting Temperature (OTC) such that IHC with difficult antibodies can be done (to potentially obtain mRNA or DNA). The IHC studies will be done at the UCSF Helen Diller Family Comprehensive Cancer Center Immunohistochemistry and Molecular Pathology Core. The tissue analyses of the biopsy and surgical specimens will be done by study pathologist.

The CT and magnetic resonance (MR) imaging analyses will be performed at the Abdominal Imaging at UCSF. To decrease the impact that metal stents may have on the functional MRI results, we will include only patients who have plastic stents in our study. In addition, to reduce variability in results, the DCE-MRI and DWI-MRI will be obtained on the same MR machine at a similar time of day as the baseline scan. The DCE-MRI images will be analyzed by calculating Ktrans and DWI-MRI images will be analyzed by calculating apparent diffusion coefficient (ADC) as described elsewhere. We will scan patients in a torso coil on a 3T clinical MR scanner. Imaging will include MR diffusion with b-values of 0, 125, and 500 for estimates of perfusion and tumor, and dynamic contrast-enhanced MR imaging (DCE-MRI) for measurement of Ktrans, blood volume, and blood flow. The region of tumor will be determined by MR imaging in reference to the baseline CT scans. The native T1 of the pancreas and liver will be calculated from a series of four, 3D, spoiled gradient recalled echo (SPGR) sequences with different flip angles. The conventional DCE-MRI will be acquired as a 3D, fast spoiled gradient echo sequence, covering the targeted areas of the pancreas or liver, at a temporal resolution of 5 sec over 6 minutes after the administration of 0.1 mmol/kg gadobenate dimeglumine. DCE-MRI images will be post-processed using MIStar software (Apollo Medical Imaging, Melbourne, Australia), which allows for motion correction to account for any shifts in data. Datasets with artifacts will be eliminated before further post processing. After contrast delivery, the new T1 is calculated and is presumed to change with the Gd concentration such that [Gd] = (1/T1-1/T10)/R1 where R1 is assumed to be 4.5 sec-1 mmol/L-1 at 3T.

Run-in Period with PEGPH20

- Days 1, 4

PEGPH20 3 ug/kg Dexamethasone 8mg PO 1-2 hours pre-PEGPH20 and PO 8-to-12 hours post-PEGPH20

*Start enoxaparin 1 mg/kg subcutaneous daily on day 1 (to be continued throughout the trial)

- On day 8 of run-in period with PEGPH20, EUS-directed core biopsy, CA 19-9, functional MRI and CT chest, abdomen (pancreatic protocol) and pelvis will be obtained.

Cycle 1 and onward

-Day 1, 8, 15

PEGPH20 3 ug/kg + Gemcitabine 1000mg/m2 + nab-Paclitaxel 125mg/m2 Dexamethasone 8mg PO 1-2 hours pre-PEGPH20 and PO 8-to-12 hours post-PEGPH20

* Gemcitabine and nab-paclitaxel will be administered 2-4 hours post-PEGPH20.
* Neoadjuvant therapy will be four 28-day cycles with CT chest, abdomen and pelvis scans and CA 19-9 measurements every 8 weeks. Patients will be taken off of the study if there is any evidence of disease progression.
* After four cycles of neoadjuvant therapy, patients will be evaluated for surgical resection depending on the CT scan findings obtained on cycle 4, day 21.
* If they have resectable disease, they will have a functional MRI following the restaging CT scan. If patients have successful resection, they will receive 2 additional cycles of gemcitabine and nab-paclitaxel. If they are found to have unresectable disease in the operating room, an intra-operative core biopsy will be obtained.
* If they have unresectable disease on the restaging scans following 4 cycles of therapy, they will be taken off of the study.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Histologically confirmed pancreatic adenocarcinoma
* Borderline resectable disease
* Performance status of Eastern Cooperative Oncology Group (ECOG) of 0-1
* Therapy naïve
* Evaluable disease with either:
* RECIST-defined measurable disease
* An elevated serum CA19-9 >100 u/ml
* Adequate organ function including:
* Bone marrow: Absolute Neutrophil Count (ANC) ≥1500/mm3, platelets ≥100,000/mm3 and hemoglobin ≥ 9 g/dL
* Hepatic: Serum total bilirubin ≤1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) and aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2.5 x ULN.
* Renal: Serum creatinine (sCr) ≤ 1.5 x ULN, or creatinine clearance (Ccr) ≥ 40 mL/min as calculated by the Modified Cockcroft-Gault formula.
* Peripheral neuropathy < grade 2
* Alkaline phosphatase ≤ 2 times the ULN unless bone metastasis is present in the absence of liver metastasis

Exclusion Criteria:

* Age younger than 18 years old
* Locally advanced or metastatic disease
* Known allergy to hyaluronidase
* Contraindications to prophylactic dose low molecular weight heparin (LMWH) , including
* Patients with recent gastrointestinal bleeding
* History of heparin induce thrombocytopenia on LMWH
* Subjects with previous severe hemorrhagic events on LMWH
* Known contraindications to heparin including:
* Recent central nervous system bleed, intracranial or spinal lesion at high risk for bleeding
* Active bleeding (major): more than 2 units transfused in 24 hours
* Spinal anesthesia/lumbar puncture within the past month
* Chronic, clinically significant measurable bleeding > 48 hours
* Severe platelet dysfunction (uremia, medications, dysplastic hematopoiesis)
* Recent major operation at high risk for bleeding
* Underlying hemorrhagic coagulopathy High risk for falls (head trauma)
* Presence of metal biliary stents (plastic biliary stents are not an exclusion)
* Known status of HIV which is not well-controlled at the time of study eligibility
* Untreated Hepatitis B infection
* Active infection or antibiotics within 48 hours prior to study
* Currently active second primary malignancy or history of malignancy less than 5 years prior to the time of study eligibility (Patients with history of skin cancers excluding melanoma will be eligible for participation).
* Serious medical comorbidities such as New York Heart Association Class III/IV cardiac disease, uncontrolled cardiac arrhythmias, myocardial infarction over the past 12 months.
* Patients with aneurysm clips, ear implants, spinal nerve stimulators, pacemaker, shrapnel or any other metal in their body (contraindication for MRI scans)
* Known, existing uncontrolled coagulopathy. Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation are eligible IF: they are appropriately anticoagulated and have not had a Grade 2 or greater bleeding episode in the 3 weeks before Day 1.
* Current use of warfarin (patients will be eligible if warfarin is discontinued and low-molecular weight heparin is used instead).
* Intolerance to dexamethasone
* Prior history of cerebrovascular accident or transient ischemic attack, or pre-existing carotid artery disease.
* Known pregnancy, nursing women or positive pregnancy test.
* Any condition that would preclude informed consent, consistent follow-up and compliance for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated earlier than expected due to low accrual so no participants were enrolled in the "Combination therapy alone" treatment arm.
Groups:
- Combination Therapy With 1 Week Run-In: PEGPH20: 3ug/kg on Days 1 and 4
  1 cycle = 28 days
  PEGPH20: 3ug/kg on Days 1, 8, 15
  Gemcitabine: 1000mg/m^2 on Days 1, 8, 15
  Nab-paclitaxel: 125mg/m^2 on Days 1, 8, 15
  PEGPH20
  Gemcitabine
  Nab-paclitaxel
- Combination Therapy Alone: 1 cycle = 28 days
  PEGPH20: 3ug/kg on Days 1, 8, 15
  Gemcitabine: 1000mg/m^2 on Days 1, 8, 15
  Nab-paclitaxel: 125mg/m^2 on Days 1, 8, 15
  PEGPH20
  Gemcitabine
  Nab-paclitaxel
Period: Overall Study
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated prior to enrollment in arm without run-in period (Combination therapy alone)
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 1 |  | 1
  70-79 years old | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinically Relevant Pancreatic Fistula
Description: Our study will be investigating only clinically relevant pancreatic fistulas, i.e. grades B or C. Descriptive statistics will be used report the incidence of pancreatic fistula within the 7-day post-operative period after neoadjuvant treatment
Time Frame: Up to 5 years
Population: No data was collected for these patients.
Groups:
- Combination Therapy Alone: 1 cycle = 28 days
  PEGPH20: 3ug/kg on Days 1, 8, 15
  Gemcitabine: 1000mg/m^2 on Days 1, 8, 15
  Nab-paclitaxel: 125mg/m^2 on Days 1, 8, 15
  PEGPH20
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Rate of Pathologic Complete Response (pCR)
Description: Descriptive statistics with frequency / proportion will be used to evaluate rate of pathologic complete response using the pathological exam of resected tumors. pCR was defined as area of scarring in pancreatic parenchyma and/or peripancreatic soft tissue with chronic inflammation, with or without acellular mucin pools and histiocytic infiltrates, but no residual viable invasive adenocarcinoma cells in the pancreatectomy specimen
Time Frame: Up to 5 years
Population: No data was collected for these patients.
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change of CA19-9 Response Rate
Description: To evaluate the disease response to treatment, CA19-9 levels will be measured every 4 weeks and restaging Computerized tomography (CT) / magnetic resonance imaging (MRI)of the chest, abdomen and pelvis will be obtained every 8 weeks
Time Frame: Up to 5 years
Population: No data was collected for this endpoint
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Margin-Negative (R0) Resection Rate
Description: Patients will be evaluated for surgical resection depending on imaging obtained on Cycle 4 Day 21. R0 Resection rate determined by CA 19-9 levels will be checked every 4 weeks and restaging CT/MRI of the chest, abdomen and pelvis will be obtained every 8 weeks surgical resection if the patient's tumor is deemed resectable post-therapy. Patients who have received at least 2 complete, 28-day cycles of study drugs were included in the secondary analyses
Time Frame: Up to 5 years
Population: No data was collected for these patients.
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Descriptive statistics with frequency and proportion of overall response determined by CA 19-9 levels will be checked every 4 weeks and restaging CT/MRI of the chest, abdomen and pelvis will be obtained every 8 weeks
Time Frame: Up to 5 years
Population: No data was collected for these patients.
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Disease Free Survival (DFS)
Description: Kaplan-Meier methods will be used to analyze disease free survival and median time and 95% confidence intervals will be reported
Time Frame: Up to 5 years
Population: No data was collected for these patients.
Arm/Group | Combination Therapy With 1 Week Run-In | Combination Therapy Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Investigator and the study team will record any occurrences of Adverse Events (AEs) from the signing of the informed consent to 28 days after the last dose of study drug, or longer if the PI deems the event is related to the drug - up to 5 years
Description: All eligible patients who are enrolled into the study and receive at least one complete, 28-day cycle of the study drugs will be included in the safety analysis. Enrollment was terminated early due to low accrual, with no patients enrolled in the combination therapy alone arm.
Arm/Group | Combination Therapy With 1 Week Run-In
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy With 1 Week Run-In (N=3)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy With 1 Week Run-In (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (8)
Edema limbs (General disorders) | 3 (7)
Fatigue (General disorders) | 3 (6)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (5)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Platelet count decreased (Investigations) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (5)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated earlier than expected due to low accrual so no participants were enrolled in the "Combination therapy alone" treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02487277/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT02487277/ICF_001.pdf